CLINICAL TRIAL: NCT06162013
Title: The NADAPT Study: a Randomized Double-blind Trial of NAD Replenishment Therapy for Atypical Parkinsonism
Acronym: NADAPT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Oslo University Hospital (Other); Akershus Universitetssykehus HF (Unknown); Vestre Viken Hospital Trust (Other); Sykehuset Ostfold (Other); Nevro Arendal AS (Unknown); Helse Forde (Other); Helse Fonna (Other); Universitetssykehuset Nord Norge HF (Unknown); Helse Møre og Romsdal HF (Other Government); Nordlandssykehuset HF (Other); Elysium Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023/634814; 2023/634814 (Other: REK Vest)
Record Dates: First submitted 2023-11-17; First posted 2023-12-08 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-10

CONDITIONS: Progressive Supranuclear Palsy; Multiple System Atrophy; Corticobasal Syndrome
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Multiple System Atrophy; Corticobasal Degeneration | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: 130 patients with PSP, 165 patients with MSA, and an undetermined number of patients with CBS will be stratified into cohorts by disease and randomized 1:1 per disease to receive either 3000mg NR a day or placebo (Fig 1). Follow up will be 18 months and consist of both in-clinic visits and decentralized patient-reported outcomes. NADAPT follows a basket trial design with parallel cohorts, essentially encompassing three trials in one, and drawing added value from the parallel enrolment and follow up.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Following our basket trial design, there will be three parallel intervention cohorts (one per disease/cohort)
  Interventions: Dietary Supplement: Nicotinamide Riboside
- Placebo (Placebo Comparator): Following our basket trial design, there will be three parallel placebo cohorts (one per disease/cohort)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — Nicotinamide Riboside 3000mg/day
  Other Names: NR
  Arms: Intervention
Other: Placebo — Placebo. Identical in taste and appearance as the intervention.
  Arms: Placebo

SUMMARY:
Progressive supranuclear palsy (PSP), Multiple system atrophy (MSA) and corticobasal syndrome (CBS) are severe neurodegenerative diseases with rapid progression and no effective treatment. Patients quickly succumb to increasing motor and non-motor symptoms and survival ranges from ~3 years to ~10 years.

Although PSP, MSA and CBS are rare diseases they constitute a major and mostly unaddressed challenge to health-care providers due to the severity of disease and lack of treatment.

The main hypothesis for the NADAPT trial is that oral administration of NR can boost cellular NAD levels in the central nervous system of patients with PSP, MSA and CBS, and rectify metabolism and inhibit neurodegeneration, resulting in delayed disease progression and amelioration of symptoms for these patients.

To test whether NR is a neuroprotective therapy for atypical parkinsonism, the investigators will perform the NADAPT clinical trial. The investigators will include 130 patients with Progressive supranuclear palsy (PSP), 165 patients with Multiple system atrophy (MSA) and an indeterminate number of patients with corticobasal syndrome (CBS). The participants will be stratified by disease into three cohorts and randomized to either 3000mg NR daily or placebo.

The trial will include patients from all of Norway. Patients will be followed for 78 weeks with both in-clinic visits and decentralized safety measurements and reporting of patient reported outcomes (PROMs). After completion of the 78 weeks follow-up, patients are offered to continue in an open-label NR-only extension study, this extension study will last until follow-up is completed for the last patients in NADAPT.

DETAILED DESCRIPTION:
Background/Rationale: Atypical parkinsonian syndromes (APS) are rapidly progressive, debilitating, and incurable neurodegenerative diseases, including progressive supranuclear palsy (PSP), multiple system atrophy (MSA) and corticobasal syndrome (CBS). These are classified as rare and orphan disorders according to EU regulation, with a reported prevalence of 7/100,000 for PSP, 4.4/100,000 for MSA, and 0.6-1/100,000 for CBS, although accurate numbers for CBS are lacking. Currently, there are no neuroprotective therapies able to delay the progression of APS. Moreover, unlike Parkinson's disease (PD), symptomatic therapy is largely ineffective. Without options for disease modification or symptom relief, patients succumb to rapidly increasing motor and cognitive disability, and become quickly care-dependent, with an estimated overall survival from diagnosis between 3-8 years for PSP, 6-10 years for MSA and ~7 years for CBS. Despite being a source of morbidity and mortality comparable to amyotrophic lateral sclerosis (ALS), there are currently no clinical treatment studies on PSP, MSA, or CBS in Norway, and very few initiatives globally. Given the complete lack of therapy - neuroprotective, symptomatic or palliative - these disorders constitute an important and urgent challenge to health care and society.

Taken together, the findings of our NAD-replenishment trials, NADPARK (NCT03816020) and NR-SAFE (NCT05344404), provide robust experimental evidence that: 1) NR has a dose-dependent symptomatic antiparkinsonistic effect, which occurs on the top of optimal dopaminergic therapy; 2) Nominate NR as a potential neuroprotective therapy for parkinsonism, able to ameliorate cerebral metabolism and dampen neuroinflammation.

Encouraged by these findings, the investigators proposed that NAD-replenishment therapy via oral NR intake could show promise as both symptomatic and neuroprotective therapy for APS. Given the complete lack of treatment options for individuals with PSP, this trial is both timely and necessary.

The investigators will conduct the NADAPT trial, a randomized, double blinded, phase II trial testing the efficacy of NAD replenishment therapy with nicotinamide riboside (NR) as a disease modifying therapy for APS. 130 patients with PSP, 165 patients with MSA, and an undetermined number of patients with CBS will be stratified by disease and randomized 1:1 per disease to receive either 3000mg NR a day or placebo (Fig 1). Follow up will be 18 months and consist of both in-clinic visits and decentralized patient-reported outcomes. NADAPT follows a basket trial design, essentially encompassing three trials in one, and drawing added value from the parallel enrolment and follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must understand the nature of the study and be able to provide written, informed consent.
2. Male or female aged 30-85 years at baseline.
3. 123I-Ioflupane dopamine transporter imaging (DaTSCAN) or FDOPA- PET has been performed. A negative DaTSCAN cannot be more than two years old at baseline.
4. Meet the MDS criteria for possible or probable PSP; or
5. Meet the MDS criteria for clinically possible or probable MSA; or
6. Meet the consensus criteria for probable or possible CBS.
7. A baseline PSPRS score of <40 for PSP, or baseline UMSARS score < 3 on items: 1, 2, 7-9.
8. Score ≥ 20 on the Mini-Mental State Examination (MMSE) at screening.
9. Able to ambulate independently or with assistance defined as the ability to take at least 5 steps with a walker (guarding is allowed provided there is no contact) or the ability to take at least 5 steps with the assistance of another person who can only have contact with one upper extremity.

Exclusion Criteria:

1. Insufficient fluency in local language to complete neuropsychological and functional assessments.
2. Evidence of differential diagnoses to PSP, MSA or CBS including: PD; dementia with Lewy bodies; Alzheimer's disease; motor neuron disease; history of repeated and/or major stroke; history of repeated and/or severe brain or spinal cord; history of neuroleptic use (except quetiapine) for prolonged period within the last 6 months; history of severe encephalitis; street drug-related parkinsonism; vascular parkinsonism; familial PSP, FTD, or known pathogenic MAPT mutation; prion disease; other neurological disease or MRI findings that could explain the PSP, MSA or CBS symptoms.
3. Presence of other significant neurological or psychiatric disorders including (but not limited to) psychotic disorders; severe bipolar or unipolar depression; seizure disorder; tumor or other space-occupying lesion.
4. Treatment with/use of NR or any investigational drugs or device, within 90 days of screening.
5. A history of alcohol or substance abuse within 1 year prior to baseline (Visit 1) and deemed to be clinically significant by the site investigator
6. Any active neoplastic malignancy (other than non-metastatic dermatological conditions) within two years of the screening visit (Visit 0) or current clinically significant hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal, or neurological disease. Active neoplastic malignancy is defined as having a known malignant focus and/or receiving anti-cancer treatment. For the non-cancer conditions, if the condition has been stable for at least the one year before the screening visit (Visit 0) and/or is judged by the site investigator not to interfere with the subject's participation in the study, the subject may be included.
7. Clinically significant laboratory abnormalities at screening that cannot be corrected to baseline and that is deemed incompatible with study participation by investigator.
8. History of deep brain stimulator surgery other than sham surgery for deep brain stimulation (DBS) clinical trial.
9. History of a clinically significant medical condition that would interfere with the subject's ability to comply with study instructions, would place the subject at increased risk, or might confound the interpretation of the study results.
10. Severe dysphagia with inability to swallow study-drug safely at baseline.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
PSP Cohort: Between group difference in PSP Rating Scale (PSPRS) total score from baseline to week 78 | 78 weeks
  Our primary outcome measure for the PSP Cohort is the between group (placebo or NR) difference in Progressive Supranuclear Palsy Rating Scale (PSPRS) total score from baseline to week 78.
MSA Cohort: Between group difference in Unified MSA Rating Scale (UMSARS) total score from baseline to week 78 | 78 weeks
  Our primary outcome measure for the MSA Cohort is the between group (placebo or NR) difference in the Unified Multiple System Atrophy Rating Scale (UMSARS) total score from baseline to week 78.
CBS Cohort: Between group difference in PSP Rating Scale (PSPRS) total score from baseline to week 78 | 78 weeks
  Our primary outcome measure for the CBS Cohort is the between group (placebo or NR) difference in Progressive Supranuclear Palsy Rating Scale (PSPRS) total score from baseline to week 78.

SECONDARY OUTCOMES:
Safety and tolerability | 79 weeks (Trial duration of 78 weeks plus 7 days after last dose of intervention or placebo)
  Monitor frequency and severity of adverse events (AE)
Specific motor/non-motor symptoms, activities of daily function, and quality of life as measured by the PSPRS | 78 weeks
  Measured by individual items of the PSPRS
Specific motor/non-motor symptoms, activities of daily function, and quality of life as measured by the UMSARS | 78 weeks
  Measured by individual items of the UMSARS
Specific motor/non-motor symptoms, activities of daily function, and quality of life as measured by the UPDRS | 78 weeks
  Measured by individual items of the Movement disorders society unified parkinson's disease rating scale (UPDRS)
Specific motor/non-motor symptoms, activities of daily function, and quality of life as measured by the MoCA | 78 weeks
  Measured by individual items of the Montreal Cognitive Assesment (MoCA)
Specific motor/non-motor symptoms, activities of daily function, and quality of life as measured by the SEADL | 78 weeks
  Measured by individual items of the Schwab and England Activities of Daily Living (SEADL)
Specific motor/non-motor symptoms, activities of daily function, and quality of life as measured by the PSP-QoL | 78 weeks
  Measured by individual items of the PSP Quality of Life questionnaire (PSP-QoL)
Specific motor/non-motor symptoms, activities of daily function, and quality of life as measured by the MSA-QoL | 78 weeks
  Measured by individual items of the MSA Quality of Life questionnaire (MSA-QoL)
Nigrostriatal degeneration | 78 weeks
  DaTSCAN tracer uptake in the striatum (total and anatomical parts).

OTHER OUTCOMES:
Daily function | 78 weeks
  Real-time wearable sensor-based data to evaluate symptoms of disease/disease burden in the home.
Brain atrophy | 78 weeks
  MRI-volumetric measurements in the frontal lobe, third ventricle, superior cerebellar peduncle, midbrain, brainstem, and whole brain.
Brain NAD metabolism | 78 weeks
  NAD levels in the brain parenchyma measured by 31P-MRS, and NAD metabolome in CSF.
Markers of neuroinflammation | 78 weeks
  Levels of selected inflammatory cytokines in serum and CSF.
CSF and serum biomarkers | 78 weeks
  Levels of amyloid beta peptide (Aβ 1-42)
CSF and serum biomarkers | 78 weeks
  Levels of tau and phosphorylated tau (PH-tau)
CSF and serum biomarkers | 78 weeks
  Levels of Neurogranin (NGRN)
CSF and serum biomarkers | 78 weeks
  Levels of neurofilament light (NfL)
CSF and serum biomarkers | 78 weeks
  Levels of neurofilament phosphorylated heavy subunit (pNfH)
Blood transcriptome. | 78 weeks
  Gene expression analyses in blood using RNA-sequencing
Blood proteome. | 78 weeks
  Proteomics in blood and/or cerebrospinal fluid using mass spectrometry
Blood metabolome. | 78 weeks
  Metabolomics in blood and/or cerebrospinal fluid using Liquid chromatography-mass spectrometry
Affects brain metabolic patterns | 78 weeks
  Measured by FDG-PET in a subset of patients (30 per cohort).

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Tzoulis, MD, PhD, Study Director — Haukeland University Hospital
Locations (3):
- Norway (3):
  - Oslo University Hospital, Oslo, Oslo County
  - Haukeland University Hospital, Bergen, Vestland
  - Vestre Viken HF, Drammen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website (Norwegian only) — https://www.helse-bergen.no/kliniske-studier/nadapt-studien/